CLINICAL TRIAL: NCT00677014
Title: SMARTDELAY Determined AV Optimization: A Comparison to Other AV Delay Methods Used in Cardiac Resynchronization Therapy
Brief Title: Comparison of AV Optimization Methods Used in Cardiac Resynchronization Therapy (CRT)
Acronym: SMART-AV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-CA-050508-H
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Results first posted 2012-08-30 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; HF; Cardiac Resynchronization Therapy; CRT; Optimization; SmartDelay; Echocardiography; AV Delay
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Echo optimized AV delay (Active Comparator): Echo optimized AV delay
  Interventions: Device: AV Delay programming through cardiac resynchronization therapy
- Algorithm optimized AV delay (Active Comparator): Algorithm optimized AV delay
  Interventions: Device: AV Delay programming through cardiac resynchronization therapy
- Fixed AV Delay (Active Comparator): Fixed AV Delay
  Interventions: Device: AV Delay programming through cardiac resynchronization therapy

INTERVENTIONS:
Device: AV Delay programming through cardiac resynchronization therapy — All subjects in this trial receive the same device. For the purpose of this trial. "intervention" is programming of the atrio-ventricular (AV) delay in the two treatment arms, while the control arm will receive AV delay programming from a Fixed nominal setting. Echo optimized and Algorithm optimized are the treatment arms programmed to receive optimized AV delay settings and will be compared to the Fixed nominal arm.
  Arms: Fixed AV Delay
Device: AV Delay programming through cardiac resynchronization therapy — All subjects in this trial receive the same device. For the purpose of this trial. "intervention" is programming of the atrio-ventricular (AV) delay in the two treatment arms, while the control arm will receive AV delay programming from a Fixed nominal setting. Echo optimized and Algorithm optimized are the treatment arms programmed to receive optimized AV delay settings and will be compared to the Fixed nominal arm.
  Arms: Algorithm optimized AV delay
Device: AV Delay programming through cardiac resynchronization therapy — All subjects in this trial receive the same device. For the purpose of this trial. "intervention" is programming of the atrio-ventricular (AV) delay in the two treatment arms, while the control arm will receive AV delay programming from a Fixed nominal setting. Echo optimized and Algorithm optimized are the treatment arms programmed to receive optimized AV delay settings and will be compared to the Fixed nominal arm.
  Arms: Echo optimized AV delay

SUMMARY:
The primary objective of SMART-AV is to assess the effect of SmartDelay for determining optimal AV delay timing during CRT compared to both a fixed AV delay and echocardiography-determined optimal AV timing chronically over a 6-month period.

DETAILED DESCRIPTION:
SMART-AV is a randomized, multi-center, double-blinded, non-significant risk, three-armed trial that will investigate the effects of optimizing AV delay timing in heart failure patients receiving CRT-D therapy. Patients will be randomized in a 1:1:1 ratio using randomly permuted blocks within each center. The study will compare chronic changes in structural and functional outcomes in CRT-D patients randomized to AV delay set as fixed, set with SmartDelay or determined by echocardiography. Patients will be followed at enrollment, implant, post-implant, 3-months post-implant and 6-months post-implant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet current indications for a BSC CRT-D device with the SmartDelay algorithm
* Patients who are willing and capable of undergoing a device implant and participating in all testing associated with the SMART-AV Study
* Patients who are on optimal and stable pharmacologic therapy
* Patients who are expected to be in sinus rhythm at the time of implant
* Patients who have a life expectancy of more than 360 days, per physician's discretion
* Patients who are geographically stable and willing to comply with the required follow-up schedule
* Patients who are 18 years of age or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

* Patients who are in complete heart block, or who otherwise are unable to tolerate pacing at VVI-40 RV for up to 14 days
* Patients undergoing an upgrade of a pacemaker or implantable cardioverter-defibrillator who are unable to tolerate pacing at VVI-40 RV for up to 14 days
* Patients who have previously received cardiac resynchronization therapy
* Patients who are expected to receive a heart transplant or have other cardiac surgeries or procedures planned during the course of the study
* Patients who currently have or who are likely to receive a tricuspid valve prosthesis
* Patients who have a neuromuscular, orthopedic, or other non-cardiac condition that prevents normal, unsupported walking
* Patients who are pregnant or planning to become pregnant during the study
* Patients who are currently enrolled in another investigational study or registry that would directly impact the treatment or outcome of the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Actual)
Dates: Start 2008-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CRM Clinical Affairs, Study Director — Boston Scientific Corporation
Locations (1):
- Medical College of Virginia, Richmond, Virginia, United States

REFERENCES:
- [Background] Auricchio A, Stellbrink C, Block M, Sack S, Vogt J, Bakker P, Klein H, Kramer A, Ding J, Salo R, Tockman B, Pochet T, Spinelli J. Effect of pacing chamber and atrioventricular delay on acute systolic function of paced patients with congestive heart failure. The Pacing Therapies for Congestive Heart Failure Study Group. The Guidant Congestive Heart Failure Research Group. Circulation. 1999 Jun 15;99(23):2993-3001. doi: 10.1161/01.cir.99.23.2993. PMID 10368116
- [Background] Auricchio A, Ding J, Spinelli JC, Kramer AP, Salo RW, Hoersch W, KenKnight BH, Klein HU. Cardiac resynchronization therapy restores optimal atrioventricular mechanical timing in heart failure patients with ventricular conduction delay. J Am Coll Cardiol. 2002 Apr 3;39(7):1163-9. doi: 10.1016/s0735-1097(02)01727-8. PMID 11923041
- [Background] Inoue N, Ishikawa T, Sumita S, Nakagawa T, Kobayashi T, Matsushita K, Matsumoto K, Ohkusu Y, Taima M, Kosuge M, Uchino K, Kimura K, Umemura S. Long-term follow-up of atrioventricular delay optimization in patients with biventricular pacing. Circ J. 2005 Feb;69(2):201-4. doi: 10.1253/circj.69.201. PMID 15671613
- [Background] Meisner JS, McQueen DM, Ishida Y, Vetter HO, Bortolotti U, Strom JA, Frater RW, Peskin CS, Yellin EL. Effects of timing of atrial systole on LV filling and mitral valve closure: computer and dog studies. Am J Physiol. 1985 Sep;249(3 Pt 2):H604-19. doi: 10.1152/ajpheart.1985.249.3.H604. PMID 3839979
- [Background] Morales MA, Startari U, Panchetti L, Rossi A, Piacenti M. Atrioventricular delay optimization by doppler-derived left ventricular dP/dt improves 6-month outcome of resynchronized patients. Pacing Clin Electrophysiol. 2006 Jun;29(6):564-8. doi: 10.1111/j.1540-8159.2006.00402.x. PMID 16784420
- [Background] Steendijk P, Tulner SA, Bax JJ, Oemrawsingh PV, Bleeker GB, van Erven L, Putter H, Verwey HF, van der Wall EE, Schalij MJ. Hemodynamic effects of long-term cardiac resynchronization therapy: analysis by pressure-volume loops. Circulation. 2006 Mar 14;113(10):1295-304. doi: 10.1161/CIRCULATIONAHA.105.540435. Epub 2006 Mar 6. PMID 16520415
- [Background] Hardt SE, Yazdi SH, Bauer A, Filusch A, Korosoglou G, Hansen A, Bekeredjian R, Ehlermann P, Remppis A, Katus HA, Kuecherer HF. Immediate and chronic effects of AV-delay optimization in patients with cardiac resynchronization therapy. Int J Cardiol. 2007 Feb 14;115(3):318-25. doi: 10.1016/j.ijcard.2006.03.015. Epub 2006 Aug 7. PMID 16891011
- [Background] Tournoux FB, Alabiad C, Fan D, Chen AA, Chaput M, Heist EK, Mela T, Mansour M, Reddy V, Ruskin JN, Picard MH, Singh JP. Echocardiographic measures of acute haemodynamic response after cardiac resynchronization therapy predict long-term clinical outcome. Eur Heart J. 2007 May;28(9):1143-8. doi: 10.1093/eurheartj/ehm050. Epub 2007 Apr 21. PMID 17449877
- [Background] Vidal B, Sitges M, Marigliano A, Delgado V, Diaz-Infante E, Azqueta M, Tamborero D, Tolosana JM, Berruezo A, Perez-Villa F, Pare C, Mont L, Brugada J. Optimizing the programation of cardiac resynchronization therapy devices in patients with heart failure and left bundle branch block. Am J Cardiol. 2007 Sep 15;100(6):1002-6. doi: 10.1016/j.amjcard.2007.04.046. Epub 2007 Jul 5. PMID 17826387
- [Background] Kedia N, Ng K, Apperson-Hansen C, Wang C, Tchou P, Wilkoff BL, Grimm RA. Usefulness of atrioventricular delay optimization using Doppler assessment of mitral inflow in patients undergoing cardiac resynchronization therapy. Am J Cardiol. 2006 Sep 15;98(6):780-5. doi: 10.1016/j.amjcard.2006.04.017. Epub 2006 Jul 28. PMID 16950184
- [Derived] Howell S, Stivland TM, Stein K, Ellenbogen K, Tereshchenko LG. Response to cardiac resynchronisation therapy in men and women: a secondary analysis of the SMART-AV randomised controlled trial. BMJ Open. 2021 Oct 27;11(10):e049017. doi: 10.1136/bmjopen-2021-049017. PMID 34706949
- [Derived] Howell SJ, Stivland T, Stein K, Ellenbogen KA, Tereshchenko LG. Using Machine-Learning for Prediction of the Response to Cardiac Resynchronization Therapy: The SMART-AV Study. JACC Clin Electrophysiol. 2021 Dec;7(12):1505-1515. doi: 10.1016/j.jacep.2021.06.009. Epub 2021 Aug 25. PMID 34454883
- [Derived] Spinale FG, Meyer TE, Stolen CM, Van Eyk JE, Gold MR, Mittal S, DeSantis SM, Wold N, Beshai JF, Stein KM, Ellenbogen KA; SMART-AV Trial Investigators. Development of a biomarker panel to predict cardiac resynchronization therapy response: Results from the SMART-AV trial. Heart Rhythm. 2019 May;16(5):743-753. doi: 10.1016/j.hrthm.2018.11.026. Epub 2018 Nov 24. PMID 30476543
- See also: Sponsor website — http://www.bostonscientific.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1060 patients were enrolled. 46 patients were not implanted with a CRT-D: screening failures (27), withdrawn by physician/sponsor (15) or withdrew consent (4). 34 implanted patients were not randomized: screening failures (13), withdrawn by physician/sponsor (14), withdrew consent (4), LTFU (2), death (1), not properly randomized (3)
Groups:
- Fixed AV Delay: Patients programmed to a Fixed nominal AV delay of 120 ms with a sensed AV offset set to 0 and the LV offset set to 0
- Echo Optimized AV Delay: Echo optimized AV delay (Iterative Method), LV offset is optional
- Algorithm Optimized AV Delay: Algorithm optimized AV delay with sensed and paced AV delay recommendations and LV offset set to 0
Period: Overall Study
Arm/Group | Fixed AV Delay | Echo Optimized AV Delay | Algorithm Optimized AV Delay
Started | 325 | 323 | 332
Completed | 281 | 282 | 283
Not Completed | 44 | 41 | 49
Not completed — Lost to Follow-up | 20 | 12 | 24
Not completed — Death | 6 | 15 | 7
Not completed — Unavailable or unreadable 6 month LVESV | 18 | 14 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed AV Delay | Echo Optimized AV Delay | Algorithm Optimized AV Delay | Total
Number analyzed (Participants) | 325 | 323 | 332 | 980
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 136 | 134 | 132 | 402
  >=65 years | 189 | 189 | 200 | 578
Age Continuous [Mean (Standard Deviation); unit: years] | 66.4 (10.6) | 65.8 (11.2) | 66.1 (11.3) | 66.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 103 | 97 | 314
  Male | 211 | 220 | 235 | 666
Region of Enrollment [Number; unit: participants]
  United States | 304 | 301 | 307 | 912
  Europe | 21 | 22 | 25 | 68

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular End-systolic Volume (LVESV)
Description: Change in square root of absolute left ventricular end systolic volume from baseline to 6 month follow up
Time Frame: 6 months
Population: Availability of baseline and 6 month echocardiograms with primary endpoint values (LVESV) among randomized patients
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Fixed AV Delay | Echo Optimized AV Delay | Algorithm Optimized AV Delay
Number analyzed (Participants) | 281 | 282 | 283
ml | -15 [-41 to 6] | -19 [-45 to 6] | -21 [-45 to 6]
Statistical Analysis 1: Comparison: Fixed AV Delay vs Echo Optimized AV Delay vs Algorithm Optimized AV Delay; Gate keeping strategy utilized for Type 1 error control described in design paper - negative results observed for initial comparisons - (each at alpha = .05) between fixed and algorithm optimized AV delay and fixed and Echo optimzied AV. Results from both of these comparisons were non-significant; Test type: Superiority or Other; p = .66, ANOVA; As LVESV values were non normal by Q-Q analysis and Shapiro-Wilk test (p<.05), a square root transform was used. model adjusted for baseline LVESV; Mean Difference (Net) = -0.1

2. Secondary Outcome: Secondary Endpoints Will Include Structural and Functional Measures
Time Frame: Chronic
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from randomization through the 6-month follow-up visit. Per trial design, serious adverse events were not collected in this trial.
Description: Source vocabulary for AE coding was not used in this trial. Serious adverse events were not collected in this trial per trial design.
Arm/Group | Fixed AV Delay | Echo Optimized AV Delay | Algorithm Optimized AV Delay
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 145/325 | 145/323 | 144/332
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fixed AV Delay (N=325) | Echo Optimized AV Delay (N=323) | Algorithm Optimized AV Delay (N=332)
PG Related (Cardiac disorders) | 6 (6) | 7 (9) | 6 (6)
RA Lead Related (Cardiac disorders) | 14 (14) | 8 (8) | 7 (7)
RV Lead Related (Cardiac disorders) | 9 (9) | 11 (13) | 7 (7)
Procedure Related (Cardiac disorders) | 32 (36) | 19 (21) | 20 (23)
LV Lead Related (Cardiac disorders) | 51 (60) | 48 (57) | 36 (39)
Cardiovascular Related (Cardiac disorders) | 71 (108) | 77 (116) | 88 (132)
Death not related to any of the other Adverse Event categories (Cardiac disorders) | 5 (5) | 7 (7) | 5 (5)
Non-Cardiovascular (General disorders) | 7 (7) | 9 (9) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less